CLINICAL TRIAL: NCT01872247
Title: A Pilot Study on the Effect of Ovarian Stimulation With r-hLH/r-hFSH, r-hFSH and hMG in Reducing Apoptosis Rate in Cumulus Cells of Patients Undergoing ICSI
Brief Title: Effect of Ovarian Stimulation With r-hLH/r-hFSH,r-hFSH and hMG in Reducing Apoptosis Rate in Cumulus Cells of Patients Undergoing ICSI
Status: Completed | Type: Observational
Sponsor: Centro di Biologia della Riproduzione, Palermo, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: apoptosis2013
Record Dates: First submitted 2013-05-27; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
HP-hMG, recombinant FSH (r-hFSH) and a combination of r-hFSH/r-hLH, are commonly used for ovarian stimulation in infertile women undergoing IVF/ICSI treatments. Several publications have compared the effectiveness of these compounds, in terms of clinical outcomes.

The aim of our study is to investigate the effects of three different ovarian stimulation protocols (HP-hMG, r-hFSH and r-hFSH/r-hLH), in a pilot prospective observational study, evaluating the effects of recombinant LH and extractive hCG (with LH like activity) on the biological outcome as well as on the clinical outcome. We will use the apoptosis rate of the cumulus cell, usually discarded after oocyte collection, as molecular biomarker to assess the oocyte quality, as biological outcome. The clinical outcome was estimated measuring implantation and ongoing pregnancy rates within and between the three different ovarian stimulation protocols

DETAILED DESCRIPTION:
HP-hMG, recombinant FSH (r-hFSH) and a combination of r-hFSH/r-hLH, are commonly used for ovarian stimulation in infertile women undergoing IVF/ICSI treatments. Several publications have compared the effectiveness of these compounds, in terms of clinical outcomes . Most of the studies have been performed in women undergoing pituitary down-regulation with a GnRH agonist long protocol, focusing on the outcome after r-hFSH and HP-hMG ovarian stimulation . Two meta-analyses showed a better outcome in terms of live birth rate for HP-hMG ovarian stimulation compared to r-hFSH in the GnRH agonist long protocol. These studies mainly compare different dose regimen of the two drugs used in the same clinical population, r-hFSH and HP-hMG. Recently other two clinical randomized studies compared, in a non-inferiority design, the same dose regimen of the two drugs. The results confirmed non inferiority of the HP-hMG formulation in terms of pregnancy rate compared to the r-hFSH formulations, but significantly higher drug consumption and lower yield in oocyte recovery.

In clinical practice HP-hMG is a clinical favored treatment when LH activity is requested for the ovarian stimulation success, due to LH activity guaranteed by extractive hCG added to this formulation.

Several studies have addressed the issue of the need or convenience of adding LH activity to FSH in ovarian stimulation in IVF/ICSI-ET in order to increase clinical outcomes in IVF/ICSI cycles , but they have not been able to address the role that LH administration plays during the follicular phase of a stimulated cycle for IVF-ET under pituitary suppression. In the case of r-hFSH administration, in normo-gonadotrophic patients, low levels of endogenous LH can persist despite pituitary down-regulation with GnRH analogues. It is known that only 1% of LH receptors need to be occupied to drive adequate ovarian steroidogenesis for reproduction. But the potential benefit of additional exogenous LH supplementation in ART is still controversial .

Different meta-analyses did not demonstrate any benefit of the r-hLH supplementation in increasing clinical outcome . However, in patients of advanced age undergoing ART, likely to include a larger proportion of poor responders, the addition of r-hLH seems to be beneficial .

In a previous study, the investigators demonstrated that r-hLH supplementation during ovarian stimulation, significantly reduces apoptosis in the cumulus cells, improving oocyte competence that is necessary for adequate fertilization and the consecutive embryogenesis that ends with implantation.

Given this background, it seems appropriate to investigate the effects of three different ovarian stimulation protocols (HP-hMG, r-hFSH and r-hFSH/r-hLH), used as routine in the ovarian stimulation therapy, in a pilot prospective observational study, evaluating the effects of recombinant LH and extractive hCG (with LH like activity) on the biological outcome as well as on the clinical outcome. The apoptosis rate of the cumulus cell, usually discarded after oocyte collection, was used as molecular biomarker to assess the oocyte quality, as biological outcome. The clinical outcome was estimated measuring implantation and ongoing pregnancy rates within and between the three different ovarian stimulation protocols

ELIGIBILITY:
Inclusion Criteria:

* normal basal level of FSH (< 12 IU/mL)
* normal body mass index (BMI = kg/m2 < 28)
* poor or hyporesponse in a previous cycle according to Bologna criteria

Exclusion Criteria:

* Azoospermia
* Endometriosis
* recurrent abortion
* recurrent failures after IVF

Ages: 30 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women after 2 years of failed spontaneous conception
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
apoptosis of cumulus cell | 1 year
  The apoptosis of cumulus cells has been investigated by "in situ" fluorescent TUNEL assay. The measure of apoptosis is the percentage of apoptotic cells on the total of cells analyzed. Usually a rate less than 15% in considered normal

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Ruvolo, Biologist, Principal Investigator — Centro di Biologia della Riproduzione, Palermo, Italy
Locations (1):
- Centro di Biologia della Riproduzione, Palermo, Italy

REFERENCES:
- [Background] Carone D, Caropreso C, Vitti A, Chiappetta R. Efficacy of different gonadotropin combinations to support ovulation induction in WHO type I anovulation infertility: clinical evidences of human recombinant FSH/human recombinant LH in a 2:1 ratio and highly purified human menopausal gonadotropin stimulation protocols. J Endocrinol Invest. 2012 Dec;35(11):996-1002. doi: 10.3275/8657. Epub 2012 Oct 22. PMID 23095369
- [Result] Ruvolo G, Bosco L, Pane A, Morici G, Cittadini E, Roccheri MC. Lower apoptosis rate in human cumulus cells after administration of recombinant luteinizing hormone to women undergoing ovarian stimulation for in vitro fertilization procedures. Fertil Steril. 2007 Mar;87(3):542-6. doi: 10.1016/j.fertnstert.2006.06.059. Epub 2006 Nov 27. PMID 17126339